CLINICAL TRIAL: NCT06121427
Title: A Prospective, Observational Clinical Study to Evaluate the Incidence of Viral Hepatitis D Relapses Upon Discontinuation of Antiviral Therapy With Bulevirtide in Patients With Chronic Hepatitis D and Negative HDV RNA
Brief Title: Incidence of Viral Hepatitis D Relapses Upon Discontinuation of Bulevirtide in Patients With Chronic Hepatitis D and Negative HDV RNA
Status: Completed | Type: Observational
Sponsor: Center of target therapy (Other)
Responsible Party: Sponsor
Other Study IDs: CTT-001
Record Dates: First submitted 2023-10-18; First posted 2023-11-08 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Hepatitis D
Keywords: bulevirtide
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study will be conducted in patients with chronic co-infection with hepatitis B and D viruses, with negative PCR for HDV RNA in peripheral blood and no signs of active liver inflammation according to blood chemistry parameters, receiving background therapy with bulevirtide for more than 48 weeks and liver biopsy performed or prescribed to be performed as part of routine practice.

After the patient has signed the Informed Consent, a portion of the liver biopsy collected as part of routine practice will be sent to the laboratory for PCR testing for HDV RNA, background therapy with bulevirtide will be interrupted, and the patient will be observed in the clinic in accordance with routine medical practice, but at least once times every 4 weeks, for timely detection of relapse of the hepatitis D and initiation of antiviral therapy. Once a relapse of viral hepatitis D is determined via the PCR HDV RNA, the patient's participation in the study will be terminated.

The collected data will be analyzed to assess the probability of relapse-free over time. Separate tests will also be conducted for subgroups of patients based on covariates such as duration of previous background therapy with bulevirtide, duration of HDV suppression, use of any other concomitant antiviral therapy during bulevirtide treatment.

DETAILED DESCRIPTION:
The main goal of this study is the following:

- To assess the probability of HDV relapse-free over time after discontinuation of background therapy with bulevirtide in patients with chronic co-infection with hepatitis B and D viruses and negative PCR HDV RNA

Primary endpoint: Occurrence of hepatitis D viral relapse.

Additional objectives in this study:

* Analyze data on the time of relapse and the duration of previous background therapy with bulevirtide, the duration of the period of HDV suppression, and the use of any other concomitant antiviral therapy during the period of treatment with bulevirtide
* Analyze relapse-free patients over 96 weeks of study follow-up
* Analyze the results of qualitative PCR (positive / negative) for hepatitis D virus RNA in a liver biopsy before discontinuing bulevirtide therapy

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of the patient to participate in the study, collect and use data
* Age 18 or older
* Background therapy with bulevirtide for at least 48 weeks
* Negative qualitative PCR test for RNA of viral hepatitis D in peripheral blood before inclusion in the study
* No active liver inflammation
* Liver biopsy performed as part of routine practice (no older than 3 weeks before inclusion in the study) or prescribed biopsy to be performed before bulevirtide interruption

Exclusion Criteria:

* Liver damage not related to viral hepatitis B and D - autoimmune hepatitis, drug or alcohol liver damage, Wilson-Konovalov disease, etc.
* Co-infection with hepatitis C virus
* Patients receiving HBV and HDV therapy not in accordance with standard practice or violations of the Instructions for the medical use of the drug/s
* Moderate/severe renal/liver dysfunction
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic co-infection with hepatitis B and D viruses with negative PCR HDV RNA who meet inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Probability of HDV relapse-free over time | 96 weeks
  To assess the probability of HDV relapse-free over time discontinuation of background therapy with bulevirtide in patients with chronic co-infection with hepatitis B and D viruses and negative PCR HDV RNA

SECONDARY OUTCOMES:
Probability of HDV relapse-free over time and the duration of previous background therapy with boulevertide | 96 weeks
  Analyze the probability of HDV relapse-free over time and the duration of previous background therapy with boulevertide
Probability of HDV relapse-free over time and the duration of the period of HDV suppression | 96 weeks
  Analyze the probability of HDV relapse-free over time and the duration of the period of HDV suppression
Probability of HDV relapse-free over time and the use of any other concomitant antiviral therapy during the period of treatment with bulevirtide | 96 weeks
  Analyze the probability of HDV relapse-free over time and the use of any other concomitant antiviral therapy during the period of treatment with bulevirtide
Relapse-free patients over 96 weeks | 96 weeks
  Analyze HDV relapse-free patients over 96 weeks
Results of qualitative PCR HDV RNA in a liver biopsy | Baseline (At the time of the patient inclusion)
  Analyze the results of qualitative PCR HDV RNA (positive / negative) in a liver biopsy before discontinuing bulevirtide therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Target Therapy, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No